CLINICAL TRIAL: NCT03136692
Title: Analysis of De-identified Data From Commercially-available App Lose It!
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: FitNow Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: Lose It! data analysis
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Overweight and Obesity
Keywords: app; weight loss; diet; behavior
MeSH Terms: conditions — Overweight; Obesity; Alzheimer Disease; Weight Loss; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lose It! commercial weight loss app — Lose It! is a commercial weight loss smart phone app designed for easy caloric tracking. It provides a free mobile and web interface for users to construct an individualized weight loss plan by entering their goal weight and desired weekly weight loss. Using the user's height, current weight, gender and age, the app generates a daily caloric budget designed for the user to reach their goal. Users can then log their caloric intake, exercise, and weight to track progress toward their goal.

SUMMARY:
The study team analyzed de-identified user data provided by the commercial app Lose It!, an entity of FitNow, Inc.

DETAILED DESCRIPTION:
The study team analyzed de-identified user data collected by Lose It! for the purposes of investigating behavioral aspects of weight loss and maintenance, including engagement with the platform; user-reported data on diet, exercise, and other behaviors; data generated by Lose It! describing macronutrient or total calorie intake; periodicity of weight-related actions; user-reported demographic information; and any data from linked applications within Lose It!. All data was anonymized and exchanged as limited data sets.

ELIGIBILITY:
Inclusion Criteria:

- New app users located in the U.S. and Canada, between 18 and 80 years of age, that are overweight (25 < BMI < 30) or obese (BMI > 30), who actively used the app each month from January to May of 2016, defined as users who logged food at least 8 times during the first or second half of each month (January, February, March, April and May).

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: New app users located in the U.S. and Canada, between 18 and 80 years of age, that are overweight (25 < BMI < 30) or obese (BMI > 30), who actively used the app each month from January to May of 2016, defined as users who logged food at least 8 times during the first or second half of each month (January, February, March, April and May).
Sampling Method: Non-Probability Sample
Enrollment: 7007 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Percent body weight lost | five months
  Percent body weight lost over first five months of 2016

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hill C, Weir BW, Fuentes LW, Garcia-Alvarez A, Anouti DP, Cheskin LJ. Relationship Between Weekly Patterns of Caloric Intake and Reported Weight Loss Outcomes: Retrospective Cohort Study. JMIR Mhealth Uhealth. 2018 Apr 16;6(4):e83. doi: 10.2196/mhealth.8320. PMID 29661750